CLINICAL TRIAL: NCT01269918
Title: A Comparison of Remifentanil and Dexmedetomidine for Craniotomy Perioperative Hemodynamics and Postoperative Pain
Acronym: RemivsDex
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10-1056
Record Dates: First submitted 2010-12-22; First posted 2011-01-04 (Estimated); Results first posted 2016-12-20 (Estimated); Last update posted 2016-12-20 (Estimated); Status verified 2016-10

CONDITIONS: Adult Intracranial Tumor; Adult Solid Tumor
Keywords: Craniotomy, pain relief; Adult solid neoplasm
MeSH Terms: conditions — Brain Neoplasms | interventions — Remifentanil; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Remifentanil (Active Comparator): Remifentanil 0.08-0.15MCG/KG/MIN INFUSION THROUGHOUT PROCEDURE BASED ON HEMODYNAMICS
  Interventions: Drug: Remifentanil
- Dexmedetomidine (Active Comparator): a loading dose of dexmedetomidine was given at 0.5 to 1 micrograms/kg ideal body weight over 15 minutes, followed by an infusion at 0.2 to 0.7 micrograms/kg/hour.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Remifentanil — Remifentanil 0.08-0.15MCG/KG/MIN INFUSION THROUGHOUT PROCEDURE BASED ON HEMODYNAMICS
  Other Names: Ultiva, G187084B
  Arms: Remifentanil
Drug: Dexmedetomidine — a loading dose of dexmedetomidine was given at 0.5 to 1 micrograms/kg ideal body weight over 15 minutes, followed by an infusion at 0.2 to 0.7 micrograms/kg/hour.
  Other Names: Precedex, Dexmedetomidine Hydrochloride
  Arms: Dexmedetomidine

SUMMARY:
This will be a randomized blinded clinical trial. Patients will be randomized to receive either a remifentanil or dexmedetomidine infusion for general anesthesia. The anesthesia team will know the result of randomization at induction. Data will be gathered by research personnel who will be blinded to the anesthetic method used. Patients will be blinded to the anesthetic they receive till they are discharged from the PACU when they will have the option to be unblinded. The Data Safety and -Toxicity Committee will review all serious adverse events and toxicity reports as well as annual reviews.

DETAILED DESCRIPTION:
Anesthesia for craniotomy presents a unique challenge to the anesthesiologist. Anesthesia for neurosurgical procedures should provide optimal surgical conditions while maintaining appropriate cerebral oxygen supply and stable systemic hemodynamics. (1) It is important to prevent patient response to noxious stimuli during the procedure like pinning, drilling of the bone, opening and manipulation of the dura etc., avoid coughing and bucking during surgery and during extubation thus necessitating a deeper level of anesthesia and analgesia. At the same time it is desirable to have the patient fully awake toward the end of the surgery in order to facilitate neurologic evaluation. Management of the above presents a challenge during induction, maintenance and extubation and also during multiple critical stages of surgery Fear of the side effects of analgesic drugs frequently leads to the under-treatment of post-craniotomy pain. (2) Nevertheless, this pain continues to be commonly observed, is frequently severe, and, if unrelieved, may cause distress for the neurosurgical patient and serious complications for the operative brain. (2) There is a need for larger trials to delineate safety and efficacy of analgesic therapies with a focus on short- and long-term outcomes.

ELIGIBILITY:
Inclusion Criteria:

Patients who undergo general anesthesia for elective surgical excision of a brain tumor with following specifications:

* Age: Older than 18
* Primary and redo cases will be included
* Duration of surgery not exceeding 6 hrs.

Exclusion Criteria:

* Patient refusal
* Emergency craniotomy
* Morbid obesity
* Uncontrolled hypertension - DBP more than 110
* Cardiac conduction defects
* Patients with chronic pain.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2011-07; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shobana Rajan, MD, Principal Investigator — The Cleveland Clinic
Locations (2):
- United States (2):
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Remifentanil | Dexmedetomidine
Started | 71 | 71
Completed | 71 | 68
Not Completed | 0 | 3
Not completed — Did not receive study drug | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Remifentanil | Dexmedetomidine | Total
Number analyzed (Participants) | 71 | 68 | 139
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (14) | 56 (14) | 56 (14)
Gender [Count of Participants; unit: Participants]
  Female | 37 | 33 | 70
  Male | 34 | 35 | 69

OUTCOME MEASURES:

1. Primary Outcome: Hemodynamics
Description: Hemodynamics were defined as mean arterial pressure (MAP), measured in milimeters of mercury (mmHg). This outcome was analyzed using a repeated measures ANOVA approach. In the outcome measure data table, mean ± standard deviation MAP was reported as the aggregate mean across time points.
Time Frame: 15, 30, 45, 60, and 90 minutes after extubation.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Remifentanil | Dexmedetomidine
Number analyzed (Participants) | 71 | 68
mmHg | 98 (11) | 88 (12)
Statistical Analysis 1: Comparison: Remifentanil vs Dexmedetomidine; Dexmedetomidine versus remifentanyl on MAP collapsed over time was estimated using a 1-tailed t test from a repeated measures ANOVA model; Test type: Non-Inferiority or Equivalence — We used a noninferiority delta of 7.5 mmHg. If noninferiority was detected, we proceeded to test for superiority; p < 0.001, t-test, 1 sided; Mean Difference (Final Values) = -9, 95% CI 2-sided [-13 to -5]
Statistical Analysis 2: Comparison: Remifentanil vs Dexmedetomidine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, t-test, 1 sided; Mean Difference (Final Values) = -9, 97.5% CI 2-sided [-13 to -4]

2. Primary Outcome: Postoperative Pain
Description: Pain was measured using the visual analogue scale (VAS), where 0 is defined as no pain and 10 is defined as worst pain imaginable. This outcome was analyzed using a repeated measures ANOVA approach. In the outcome measure data table, mean ± standard deviation pain was reported as the aggregate mean across time points.
Time Frame: 15, 30, 45, 60, and 90 minutes after extubation.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Remifentanil | Dexmedetomidine
Number analyzed (Participants) | 71 | 68
units on a scale | 5.1 (2.4) | 2.9 (2.6)
Statistical Analysis 1: Comparison: Remifentanil vs Dexmedetomidine; Dexmedetomidine versus remifentanyl on VAS pain score estimated from a 1-tailed t test from a repeated measures ANOVA model; Test type: Non-Inferiority or Equivalence — We used a noninferiority delta of 1 point. If noninferiority was detected, we proceeded to test for superiority; p < 0.001, t-test, 1 sided; Mean Difference (Final Values) = -1.9, 95% CI 2-sided [-2.7 to -1.1]
Statistical Analysis 2: Comparison: Remifentanil vs Dexmedetomidine; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, t-test, 1 sided; Mean Difference (Final Values) = -1.9, 97.5% CI 2-sided [-2.8 to -0.9]

3. Primary Outcome: Total Opioid Consumption
Description: Total opioid consumption was defined as the sum of all opioid doses given within the first 90 minutes after surgery, converted to milligram morphine equivalents.
Time Frame: Initial 90 minutes of recover after surgery
Measure: Median (Inter-Quartile Range); unit: mg morphine equivalents
Arm/Group | Remifentanil | Dexmedetomidine
Number analyzed (Participants) | 71 | 68
mg morphine equivalents | 10 [7 to 15] | 5 [0 to 10]
Statistical Analysis 1: Comparison: Remifentanil vs Dexmedetomidine; Dexmedetomidine versus remifentanyl on opioid consumption estimated from a Wilcoxon rank sum test; Test type: Non-Inferiority or Equivalence — Noninferiority delta = 2 mg opioid; p < 0.001, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -5, 95% CI 2-sided [-10 to -5]
Statistical Analysis 2: Comparison: Remifentanil vs Dexmedetomidine; Dexmedetomidine versus remifentanyl on opioid consumption estimated from a Wilcoxon rank sum test; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -5, 97.5% CI 2-sided [-10 to -3]

4. Secondary Outcome: Heart Rate
Description: Heart rate was determined from the arterial catheter and measured as beats per minute. This outcome was analyzed using a repeated measures ANOVA approach.
Time Frame: 15, 30, 45, 60, and 90 minutes after extubation.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Remifentanil | Dexmedetomidine
Number analyzed (Participants) | 71 | 68
beats per minute
  Heart rate 15 minutes after extubation | 76 (15) | 68 (13)
  Heart rate 30 minutes after extubation | 72 (14) | 67 (13)
  Heart rate 45 minutes after extubation | 73 (14) | 66 (13)
  Heart rate 60 minutes after extubation | 73 (13) | 66 (12)
  Heart rate 90 minutes after extubation | 75 (13) | 69 (14)
Statistical Analysis 1: Comparison: Remifentanil vs Dexmedetomidine; Dexmedetomidine versus remifentanyl on heart rate was assessed using a linear mixed effects model adjusting for baseline heart rate; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -6, 95% CI 2-sided [-10 to 3]

5. Secondary Outcome: Modified Short Orientation Memory Concentration Test (SOMCT)
Description: The Modified Short Orientation Memory Concentration Test (SOMCT) is a validated questionnaire that discriminates among mild, moderate, and severe cognitive deficits. SOMCT is based on 6 questions and produces a total score ranging from 0 (worst possible function) to 28 (best possible function). Scores > 20 are considered normal. This outcome was analyzed using a repeated measures ANOVA approach.
Time Frame: 15, 30, 45, 60, and 90 minutes after extubation.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Remifentanil | Dexmedetomidine
Number analyzed (Participants) | 71 | 68
units on a scale
  SOMCT 15 minutes after extubation | 22 (9) | 18 (11)
  SOMCT 30 minutes after extubation | 25 (7) | 20 (11)
  SOMCT 45 minutes after extubation | 25 (6) | 23 (9)
  SOMCT 60 minutes after extubation | 26 (5) | 24 (7)
  SOMCT 90 minutes after extubation | 26 (5) | 25 (7)
Statistical Analysis 1: Comparison: Remifentanil vs Dexmedetomidine; Dexmedetomidine versus remifentanyl on SOMCT estimated using a linear mixed effects model adjusting for baseline SOMCT score; Test type: Superiority or Other; p = 0.16, Mixed Models Analysis; Mean Difference (Final Values) = -1.1, 95% CI 2-sided [-2.6 to 0.5]

6. Secondary Outcome: Aldrete Score
Description: The Aldrete score measured level of sedation and fitness and is used to assess the appropriate departure time from the post anesthesia care unit. The score ranges from 0 to 10, where 0 indicates poor fitness (and such patients are transferred to the ICU), while 10 indicates good fitness. This outcome was analyzed using a repeated measures ANOVA approach.
Time Frame: 15, 30, 45, 60, and 90 minutes after extubation.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Remifentanil | Dexmedetomidine
Number analyzed (Participants) | 71 | 68
units on a scale
  Aldrete score at 15 minutes after extubation | 8.4 (1) | 8 (1.4)
  Aldrete score at 30 minutes after extubation | 8.7 (1) | 8.3 (1.4)
  Aldrete score at 45 minutes after extubation | 9.0 (1.0) | 8.7 (1.1)
  Aldrete score at 60 minutes after extubation | 9.2 (0.9) | 8.9 (1.1)
  Aldrete score at 90 minutes after extubation | 9.4 (0.8) | 9.1 (1.1)
Statistical Analysis 1: Comparison: Remifentanil vs Dexmedetomidine; Dexmedetomidine versus remifentanyl on Aldrete score estimated using a linear mixed effects model adjusting for baseline Aldrete score; Test type: Superiority or Other; p = 0.07, Mixed Models Analysis; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-0.6 to 0.03]

7. Secondary Outcome: Nursing Workload Comparison
Description: To evaluate the nurses workload when either of the two drugs are given in terms Nursing Research Usage form's therapeutic index scoring system. This score ranges from 0 (minimal interventions and time spent by nurses on study patient) to 22 (maximum interventions and time spent by nurses on the study patient).
Time Frame: 90 minutes after extubation
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Remifentanil | Dexmedetomidine
Number analyzed (Participants) | 71 | 68
units on a scale | 6 [6 to 8] | 5.5 [5 to 7]
Statistical Analysis 1: Comparison: Remifentanil vs Dexmedetomidine; Dexmedetomidine versus remifentanyl on Nursing workload comparison estimated using a Wilcoxon rank sum test; Test type: Superiority or Other; p = 0.009, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -1, 95% CI 2-sided [-1 to -0.001]

8. Secondary Outcome: Drug Stop Time to Open Eyes
Description: time until patient first opened their eyes, squeezed a hand, or wiggled their toes in response to verbal commands after surgery
Time Frame: Anesthesia drug stop time to open eyes. Time is measured continuously until patients eyes open, regardless of how long it takes.
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Remifentanil | Dexmedetomidine
Number analyzed (Participants) | 71 | 68
minutes | 8 [7 to 9] | 38 [29 to 44]
Statistical Analysis 1: Comparison: Remifentanil vs Dexmedetomidine; Remifentanyl versus Dexmedetomidine on time to open eyes estimated using Cox regression; Test type: Superiority or Other; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 0.11, 95% CI 2-sided [0.07 to 0.18]

9. Secondary Outcome: Drug Stop Time to Recall
Description: Time between extubation until patients could say their names.
Time Frame: Time between extubation until patients could say their names.
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Remifentanil | Dexmedetomidine
Number analyzed (Participants) | 71 | 68
minutes | 13 [10 to 15] | 42 [36 to 49]
Statistical Analysis 1: Comparison: Remifentanil vs Dexmedetomidine; Remifentanyl versus dexmedetomidine on time to recall assessed using Cox regression; Test type: Superiority or Other; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 0.12, 95% CI 2-sided [0.07 to 0.19]

10. Secondary Outcome: Drug Stop Time to Fitness to Discharge
Time Frame: Anesthesia drug stop time to fitness to discharge. Time is measured continuously until fitness for discharge is reached, regardless of how long it takes.
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Remifentanil | Dexmedetomidine
Number analyzed (Participants) | 71 | 68
minutes | 150 [117 to 175] | 172 [160 to 206]
Statistical Analysis 1: Comparison: Remifentanil vs Dexmedetomidine; Remifentanyl versus Dexmedetomidine on time to fitness discharge estimated using Cox regression; Test type: Superiority or Other; p = 0.022, Regression, Cox; Hazard Ratio (HR) = 0.68, 95% CI 2-sided [0.48 to 0.95]

11. Secondary Outcome: End Case to Post Anesthesia Care Unit (PACU) Discharge
Description: Post Anesthesia Care Unit (PACU) Discharge time is the timing at which patients are discharged from the PACU. This outcome is the amount of time (minutes) from end case to PACU discharge.
Time Frame: End case to post anesthesia care unit (PACU) discharge. Time is measured continuously until PACU discharge, regardless of how long it takes.
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Remifentanil | Dexmedetomidine
Number analyzed (Participants) | 91 | 68
minutes | 211 [183 to 228] | 215 [184 to 236]
Statistical Analysis 1: Comparison: Remifentanil vs Dexmedetomidine; Remifentanyl versus Dexmedetomidine on time to PACU discharge estimated using Cox proportional hazard regression; Test type: Superiority or Other; p = 0.45, Regression, Cox; Hazard Ratio (HR) = 1.1, 95% CI 2-sided [0.81 to 1.62]

12. Secondary Outcome: Postoperative Nausea
Description: Indicator of whether patients had nausea or not
Time Frame: Whether patients had nausea or not, from anesthesia stop time until hospital discharge.
Measure: Number; unit: participants
Arm/Group | Remifentanil | Dexmedetomidine
Number analyzed (Participants) | 71 | 68
participants | 12 | 12
Statistical Analysis 1: Comparison: Remifentanil vs Dexmedetomidine; Dexmedetomidine versus remifentanyl on postoperative nausea estimated from chi squared test; Test type: Superiority or Other; p = 0.91, Chi-squared; Risk Ratio (RR) = 1.0, 95% CI 2-sided [0.5 to 2.2]

13. Secondary Outcome: Postoperative Vomitting
Description: Indicator of whether patients had postoperative vomiting.
Time Frame: Whether patients had vomiting or not, from anesthesia stop time until hospital discharge.
Measure: Number; unit: participants
Arm/Group | Remifentanil | Dexmedetomidine
Number analyzed (Participants) | 71 | 68
participants | 6 | 2
Statistical Analysis 1: Comparison: Remifentanil vs Dexmedetomidine; Dexmedetomidine versus remifentanyl on postoperative vomiting estimated from a chi square test; Test type: Superiority or Other; p = 0.16, Chi-squared; Risk Ratio (RR) = 0.4, 95% CI 2-sided [0.07 to 1.7]

14. Secondary Outcome: Postoperative Shivering
Description: Indicator of whether patients had postoperative shivering.
Time Frame: Whether patients had postoperative or not, from anesthesia stop time until hospital discharge.
Measure: Number; unit: participants
Arm/Group | Remifentanil | Dexmedetomidine
Number analyzed (Participants) | 71 | 68
participants | 7 | 3
Statistical Analysis 1: Comparison: Remifentanil vs Dexmedetomidine; Dexmedetomidine versus remifentanyl on incidence of shivering estimated from a chi square test; Test type: Superiority or Other; p = 0.21, Chi-squared; Risk Ratio (RR) = 0.4, 95% CI 2-sided [0.1 to 1.7]

ADVERSE EVENTS:
Arm/Group | Remifentanil | Dexmedetomidine
Serious Adverse Events (participants affected / at risk) | 0/71 | 0/68
Other Adverse Events (participants affected / at risk) | 0/71 | 0/68

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No